CLINICAL TRIAL: NCT06943794
Title: Gastric Cancer Prevention Strategies Based on Eradication of Helicobacter Pylori Subtypes at High Risk for Gastric Cancer: a Multicenter, Pragmatic Randomized Controlled Trial
Brief Title: Eradication of Helicobacter Pylori Subtypes at High Gastric Cancer Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Director of the gastric surgery department, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025RCT
Record Dates: First submitted 2025-03-20; First posted 2025-04-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-03

CONDITIONS: Gastric (Stomach) Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Treatment group (high-risk Hp subtype guidance + eradication treatment):
  A high-risk Hp subtype guidance group consisting of the receiving physician + trial-related personnel conducts individualized assessment based on Hp infection, SNP test results, gastric mucosa condition, medical history and other factors, and provides subjects with medical explanations and recommendations for eradication treatment.
  Eradication group protocol: standard quadruple therapy for H. pylori eradication program (PPI + bismuth + two antibiotics)
  1. Omeprazole (or esomeprazole): 20mg, 2 times/day
  2. Bismuth citrate: 220mg, 2 times/day
  3. Metronidazole: 400mg, 3 times/day
  4. Tetracycline: 500mg, 3 times/day
  5. Treatment cycle: 10-14 days Eradication success was assessed after 1 month by urea breath test (UBT) or Hp fecal antigen test.
  Follow-up:
  After 3 months: assess Hp status, recommend gastroscopy if necessary. After 1 year: review of Hp infection status, assessment of gastric mucosal lesion progression.
Who Masked: Participant
Masking Description: Subjects (high-risk SNP-positive) are uninformed about their group assignment (conventional treatment, intervention guidance) during the study. The high-risk Hp subtype steering group was informed about their subgroup. Collection of assessment data and data analysis statisticians were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (high-risk Hp subtype guidance + eradication treatment) (Experimental)
  Interventions: Drug: recommendations for eradication treatment
- Control group (routine Hp management) (No Intervention): according to the routine management of asymptomatic infected patients, will not be given the guidance intervention of high-risk Hp subtype guidance group.

INTERVENTIONS:
Drug: recommendations for eradication treatment — A high-risk Hp subtype guidance group consisting of the receiving physician + trial-related personnel conducts individualized assessment based on Hp infection, SNP test results, gastric mucosa condition, medical history and other factors, and provides subjects with medical explanations and recommendations for eradication treatment.
  Eradication group protocol: standard quadruple therapy for H. pylori eradication program (PPI + bismuth + two antibiotics)
  1. Omeprazole (or esomeprazole): 20mg, 2 times/day
  2. Bismuth citrate: 220mg, 2 times/day
  3. Metronidazole: 400mg, 3 times/day
  4. Tetracycline: 500mg, 3 times/day
  5. Treatment cycle: 10-14 days Eradication success was assessed after 1 month by urea breath test (UBT) or Hp fecal antigen test.
  Arms: Treatment group (high-risk Hp subtype guidance + eradication treatment)

SUMMARY:
This study is a prospective, multicenter randomized controlled study. Additional fecal screening for Hp-specific SNP mutation sites on top of routine Hp testing may improve the identification of people at high risk for gastric cancer, and the treatment of eradication interventions in high-risk groups can significantly reduce the incidence or risk of progression of gastric cancer.

DETAILED DESCRIPTION:
Primary study objective: To evaluate whether H. pylori eradication therapy can reduce the risk of gastric mucosal lesion progression or gastric cancer in a subgroup of asymptomatic H. pylori-positive subjects with high-risk SNP loci.

The secondary objectives of the study are: 1. to compare the difference between the "fecal Hp high-risk subtype eradication" strategy and routine Hp testing in detecting early gastric cancer or precancerous lesions (e.g., gastric mucosal atypia, intestinal metaplasia, etc.). 2. to evaluate the impact of the "fecal high-risk subtype eradication" strategy on treatment and management adherence. 3. to assess the effectiveness of the "Hp high-risk subtype eradication" strategy in reducing the risk of gastric cancer. Evaluate the impact of the "fecal high-risk Hp subtype eradication" strategy on adherence to treatment and management. 3. Analyze the improvement of gastric mucosal atrophy, intestinal metaplasia, and inflammation after eradication treatment in the "high-risk Hp subtype" population.

People meeting the inclusion criteria were recruited from multiple centers. Randomization: Subjects with high-risk subtypes who met the inclusion criteria were randomized into an intervention group and a control group. INTERVENTION: Intervention group: received standardized H. pylori eradication treatment recommendations given by trial staff/physicians based on patient risk, clinical symptoms, etc. Control group: received standardized follow-up and routine management without treatment guidance for high-risk Hp subtypes. Follow-up and comparison: to compare the differences between the two groups in terms of the detection rate of gastric cancer or precancerous lesions, the incidence (or progression) of gastric cancer, patient adherence, and complications within a certain follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Volunteer to participate in this study and sign an informed consent form.
3. Have not received H. pylori eradication treatment in the past 1 month.
4. Able to complete stool sample collection and related examinations according to the requirements of the study.
5. Have been detected as high risk by Hp subtype test.
6. Have no obvious clinical symptoms, or have mild symptoms that do not meet the current clinical guidelines for "eradication therapy".
7. Within 90 days, the gastroscopy and/or pathological results confirm the absence of gastric cancer.

Exclusion Criteria:

1. Negative Hp test.
2. Previous diagnosis of gastric cancer or other malignant tumors.
3. Severe systemic diseases or comorbidities (hepatic, renal, cardiac insufficiency, etc.) that do not tolerate gastroscopy or study procedures.
4. Use of proton pump inhibitors, antibiotics, or other drugs that affect Hp detection or therapeutic effects within 3 months.
5. Pregnant or lactating women.
6. Other conditions that the investigator considers inappropriate for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4824 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Gastric cancer-free survival in the population during follow-up. | through study completion, an average of 5 year

IPD SHARING:
Plan to Share IPD: Undecided